CLINICAL TRIAL: NCT07197385
Title: Comparison of Ureteroscopic Lithotripsy and Laparoscopic Ureterolithotomy for the Treatment of Unilateral Upper Ureteral Stone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lahore General Hospital (Other Government)
Responsible Party: Principal Investigator, Muhammad Irfan Jamil, Principal Investigator, Lahore General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LahoreGeneralH11
Record Dates: First submitted 2025-09-21; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Ureteral Calculi; Urolithiasis
Keywords: Ureteral Stones; Upper Ureteric Calculi; Ureteroscopic Lithotripsy; Ureteroscopy; Laparoscopic Ureterolithotomy
MeSH Terms: conditions — Ureteral Calculi; Urolithiasis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Laparoscopic Ureterolithotomy (LU) (Experimental): Patients randomized to this group will undergo laparoscopic ureterolithotomy under general anesthesia. Prior to the procedure, an X-ray KUB will be performed to confirm the stone location. The patient will be placed in a flank position. Pneumoperitoneum will be created using a Veress needle, and three laparoscopic ports will be placed:
  Port I (10 mm, sub-umbilical): for the 30° laparoscope
  Port II (10 mm, mid-clavicular, iliac spine level): for stone extraction
  Port III (5 mm, subcostal, mid-clavicular): for assistance and retraction
  The stone will be identified as a ureteral bulge, confirmed by palpation with an atraumatic grasper. A longitudinal ureterotomy will be performed with a laparoscopic scalpel/L-hook, and the stone will be extracted via Port II. Large stones may be placed in a gloved finger pouch for retrieval at the end of surgery. The ureterotomy will be closed with interrupted 4-0 polyglactin sutures (two or three, depending on size). A 20F Nelaton tube drain will be
  Interventions: Procedure: Laparoscopic Ureterolithotomy
- Group Ureteroscopic Lithotripsy (URS) (Active Comparator): Patients randomized to this group will undergo ureteroscopic lithotripsy under general or regional anesthesia. A cystoscopy and retrograde pyelogram will be performed first. A 6/7.5 Fr semirigid ureteroscope will be advanced through the ureteric orifice using a guidewire until the stone is visualized. Pneumatic lithotripsy will then be performed with the following settings:
  Energy: 4 bar Frequency: 5 Hz
  The stone will be fragmented into pieces <2 mm in size. A stone cone will be used to prevent retropulsion. Ureteric orifice dilatation will be performed if required. A DJ stent will be placed at the end of the procedure and will be removed at 4 weeks postoperatively. Antibiotic prophylaxis will be administered perioperatively.
  Interventions: Procedure: Ureteroscopic Lithotripsy

INTERVENTIONS:
Procedure: Laparoscopic Ureterolithotomy — Keyhole laparoscopic approach to remove proximal ureteral stones by direct ureteral incision and closure.
  Arms: Group Laparoscopic Ureterolithotomy (LU)
Procedure: Ureteroscopic Lithotripsy — Semirigid ureteroscopic fragmentation of upper ureteral stones using pneumatic lithotripsy.
  Arms: Group Ureteroscopic Lithotripsy (URS)

SUMMARY:
Kidney stones are a common health problem that can cause severe pain, blockage of urine flow, and even long-term kidney damage if left untreated. When stones move from the kidney into the upper part of the ureter (the tube that carries urine to the bladder), treatment often becomes more difficult. Several treatment options are available, including breaking the stones with sound waves, removing them with small telescopes, or performing surgery. However, the best method for larger stones in the upper ureter is still debated.

This study will compare two commonly used minimally invasive surgical techniques for removing upper ureteral stones. The first method is ureteroscopic lithotripsy (URS), in which a thin scope is passed through the urinary passage to directly reach the stone and break it into small pieces using a pneumatic device. The second method is laparoscopic ureterolithotomy (LU), a keyhole surgical procedure in which small incisions are made in the abdomen, and the stone is removed directly through the ureter.

Fifty-six adult patients with a single upper ureteral stone measuring 10-20 mm will be randomly assigned to either URS or LU. Both groups will undergo standard preoperative evaluations, and infection will be treated before surgery. The outcomes will be assessed in terms of operation time, length of hospital stay, level of postoperative pain, use of pain medications, complications during or after surgery, and the stone-free rate (absence of residual stone fragments larger than 3 mm after four weeks).

By comparing these two procedures, this study aims to identify which treatment is safer and more effective for patients with upper ureteral stones. The results will provide useful evidence to guide doctors and patients in making the best treatment choices.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders with age ≥ 18 years.
* Patients with a duration of symptoms for more than 1 month.
* Patients having a unilateral single stone of 10 mm to 20 mm in diameter, located between the ureteropelvic junction and the upper border of the sacroiliac joint (upper ureteral stone).

Exclusion Criteria:

* Patients with a history of ipsilateral ureteric surgeries, previous open abdominal surgeries, bleeding disorders and pregnancy.
* Before surgery, patients had a positive urine culture, fever (37.60c) and leukocytosis > 12.000 per microliter.
* Patients having solitary kidney and co-morbidities e.g., cardiovascular, Liver, respiratory illnesses, or serum creatinine >1.5 mg/dl.
* Horseshoe kidneys, pelvic kidneys, pyonephrosis, ureteropelvic junction blockage, and ureteral stricture.
* Patients with unsuitable for general anesthesia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2025-01-10 (Actual); Primary Completion 2025-06-10 (Actual); Study Completion 2025-06-10 (Actual)

PRIMARY OUTCOMES:
Operative Time | Intraoperative, recorded at the time of surgery
  Operative time will be measured from the start of the surgical procedure until urethral catheterization is completed. The duration will be recorded in minutes for each patient and compared between ureteroscopic lithotripsy and laparoscopic ureterolithotomy groups.
Stone-Free Rate (SFR) | At 4 weeks postoperatively (before removal of DJ stent).
  The stone-free rate will be defined as the absence of residual stone fragments >3 mm, confirmed by radiological imaging (X-ray KUB or NCCT) at follow-up. Patients with residual fragments ≤3 mm will be considered stone-free, while those with larger fragments or requiring auxiliary procedures will be considered not stone-free.

SECONDARY OUTCOMES:
Postoperative Pain (VAS Score) | Day of surgery and postoperative day 1.
  Pain intensity will be assessed using a Visual Analogue Scale (VAS) ranging from 0 (no pain) to 10 (worst pain). Scores will be recorded on the day of surgery and the first postoperative day. Analgesic use (mg dose administered) will also be documented.

CONTACTS AND LOCATIONS:
Locations (1):
- Lahore General Hospital, Lahore, Lahore, Punjab Province, Pakistan